CLINICAL TRIAL: NCT03335670
Title: Biodistribution of Ga-68 Pentixafor in Patients With Neuroendocrine Tumors
Brief Title: Gallium 68 Pentixafor in Patients With Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yusuf Menda (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Yusuf Menda, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201708705; P50CA174521 (NIH)
Record Dates: First submitted 2017-10-12; First posted 2017-11-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Tumors
Keywords: 68Ga-pentixafor; (68Ga)pentixafor; Gallium Radioisotopes; CXCR4
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 68Ga-pentixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]Pentixafor PET scan (Experimental): 4 mCi (range 3-5 mCi) of [68Ga]Pentixafor is administered intravenously over 1 minute using an infusion pump. PET imaging is performed from time of infusion for about 90 minutes. Approximately 12 blood samples (~ 1 tsp) will be taken for pharmacokinetic analysis.
  Interventions: Drug: [68Ga]Pentixafor

INTERVENTIONS:
Drug: [68Ga]Pentixafor — 68Ga Pentixafor is a radiolabeled cyclic pentapeptide with high affinity for CXCR4 receptor
  Other Names: (68Ga)pentixafor

SUMMARY:
This study will evaluate how Gallium-68 Pentixafor is distributed in neuroendocrine tumor patients and if that distribution is consistent through repeated scans. This is an RDRC study - as such, the images obtained for this study cannot be used clinically or shared with treating oncologists.

DETAILED DESCRIPTION:
High grade neuroendocrine tumors often do not express somatostatin (sstr) receptors but often express the CXCR4 receptor. The CXCR4 receptor is a marker of poorly differentiated cells. Pentixafor is a peptide that targets these CXCR4 receptors. By combining it with gallium-68, a radionuclide, pentixafor can then be evaluated as an imaging agent to detect high-grade neuroendocrine tumors.

[68Ga]Pentixafor is a radio-labelled imaging agent used for positron emission tomography (PET). The dose is small, known as a tracer dose. It is designed to capture information about the body and how the body is working without interfering or causing an effect.

The goal of this study is to evaluate how the [68Ga]Pentixafor is distributed through the body after injection and how it is taken up by the organs of the body. The study will also examine if the imaging is reproducible to determine if the PET images show the same uptake of the study drug across different scans.

This study is an RDRC study - the equivalent to a phase 0 study. The [68Ga]Pentixafor has not been shown to target tumors; specificity and sensitivity have not been established. For this reason, images obtained for this study cannot be used clinically or shared with treating oncologists.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histological diagnosis of neuroendocrine tumor (NET).
3. Had a prior 68Ga DOTATATE PET/CT scan (NetSpot) and a CT or MRI with or without contrast performed within 3 months before signing the consent, without interval treatment other than a somatostatin analog.
4. CT or MRI must demonstrate at least one lesion (primary or metastatic) present 1.5 cm or larger in any dimension on cross-sectional imaging (CT or MRI) obtained within 3 months of study enrollment.
5. Results of CXCR4 immunohistochemistry or slides from biopsy of primary tumor or metastatic lesions available for study analysis.
6. Participation in the Iowa Neuroendocrine Tumor Registry.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring hospitalization, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Physical limitation that would limit compliance with the study requirements
3. Pregnant or lactating women. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A negative pregnancy test will be required for all female subjects with child bearing potential.
4. Planned administration of any NET therapy between scan 1 and 2, except for Somatostatin analog.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Determine biodistribution (pharmacokinetic parameters) of [68Ga]Pentixafor in patients with neuroendocrine tumors (NETs) | Within 1 month of [68Ga]Pentixafor scan
  Biodistribution will be assessed through the radiotracer parameters standardized uptake value (SUV) and K-influx obtained from PET scan and blood samples.These values provide a pharmacokinetic profile of the investigational drug's biodistribution in the body.
Determine the repeatability of [68Ga]Pentixafor uptake in known neuroendocrine tumor lesions | Within 1 month of the second [68Ga]Pentixafor scan
  Determine the difference, in any, of the biodistribution values between scans 1 and 2, for subjects who undergo 2 [68Ga]Pentixafor scans.

SECONDARY OUTCOMES:
Compare standardized uptake values of [68Ga]Pentixafor and [68Ga]DOTATATE in known neuroendocrine tumor lesions | Within 6 months of [68Ga]Pentixafor scan
  The standardized uptake value (SUV) of known neuroendocrine tumors for the investigational agent [68Ga]Pentixafor will be compared to the SUV for [68Ga]DOTATATE (NetSpot).
Correlate the uptake of [68Ga]Pentixafor and [68Ga]DOTATATE (NetSpot) in known neuroendocrine tumor lesions with expression of receptors (CXCR4 and SSTR2) in biopsy tissue samples. | Within 6 months of [68Ga]Pentixafor scan
  The standardized uptake value (SUV) of the gallium PET tracers ( [68Ga]Pentixafor and/or [68Ga]DOTATATE) will be compared to the receptor expression score (H-score)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, MD, Principal Investigator — University of Iowa; M. Sue O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request to the study's principal investigator. A signed usage agreement will need to be provided.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the study has been completed.
Access Criteria: Individual participant data will be shared upon request to the study's principal investigator. A signed usage agreement will need to be provided.

REFERENCES:
- [Background] Lapa C, Luckerath K, Kleinlein I, Monoranu CM, Linsenmann T, Kessler AF, Rudelius M, Kropf S, Buck AK, Ernestus RI, Wester HJ, Lohr M, Herrmann K. (68)Ga-Pentixafor-PET/CT for Imaging of Chemokine Receptor 4 Expression in Glioblastoma. Theranostics. 2016 Jan 25;6(3):428-34. doi: 10.7150/thno.13986. eCollection 2016. PMID 26909116
- [Background] Bluemel C, Hahner S, Heinze B, Fassnacht M, Kroiss M, Bley TA, Wester HJ, Kropf S, Lapa C, Schirbel A, Buck AK, Herrmann K. Investigating the Chemokine Receptor 4 as Potential Theranostic Target in Adrenocortical Cancer Patients. Clin Nucl Med. 2017 Jan;42(1):e29-e34. doi: 10.1097/RLU.0000000000001435. PMID 27819856
- [Background] Herhaus P, Habringer S, Philipp-Abbrederis K, Vag T, Gerngross C, Schottelius M, Slotta-Huspenina J, Steiger K, Altmann T, Weisser T, Steidle S, Schick M, Jacobs L, Slawska J, Muller-Thomas C, Verbeek M, Subklewe M, Peschel C, Wester HJ, Schwaiger M, Gotze K, Keller U. Targeted positron emission tomography imaging of CXCR4 expression in patients with acute myeloid leukemia. Haematologica. 2016 Aug;101(8):932-40. doi: 10.3324/haematol.2016.142976. Epub 2016 May 12. PMID 27175029